CLINICAL TRIAL: NCT00698529
Title: Communication Technology to Disseminate Evidence-Based HIV Interventions to NGOs
Brief Title: Effectiveness of Communication Technology in Disseminating HIV Prevention Training to Non-governmental Organizations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Kelly, Professor of Psychiatry and Behavioral Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH079730 (NIH); R01MH079730 (NIH); DAHBR 9A-ASPQ
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: HIV Infections
Keywords: Technology Transfer; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Patient Portals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No POL Training (No Intervention): Participating NGOs and their staff will receive no specialized training.
- Face-to-Face (Experimental): Participating NGOs and their staff will receive training through face-to-face seminars held at the NGOs and through post-seminar consultation telephone calls.
  Interventions: Behavioral: Face-to-face training; Behavioral: Popular Opinion Leader (POL)
- Distance Learning (Experimental): Participating NGOs and their staff will receive training through Web-based seminars and through post-seminar consultation telephone calls.
  Interventions: Behavioral: Distance training; Behavioral: Popular Opinion Leader (POL)

INTERVENTIONS:
Behavioral: Face-to-face training — NGOs will receive the POL intervention through face-to-face training. Staff will receive 2-day training on the POL intervention and individualized telephone follow-up consultations concerning POL implementation.
  Other Names: Traditional; Seminar
  Arms: Face-to-Face
Behavioral: Distance training — NGOs will receive the POL intervention through Web-based training. Staff will receive training delivered entirely by means of a Web-based, distance learning curriculum and through individualized telephone follow-up consultations concerning POL implementation.
  Other Names: On-line; Internet; Distance learning
  Arms: Distance Learning
Behavioral: Popular Opinion Leader (POL) — POL is a community-level HIV intervention that recruits and trains opinion leaders in the community to promote safe sex behaviors through risk-reduction conversations with peers.
  Arms: Distance Learning; Face-to-Face

SUMMARY:
This study will compare the effectiveness of face-to-face training versus Web-based training seminars in disseminating HIV prevention interventions to nongovernmental organizations in Eastern Europe and Central Asia.

DETAILED DESCRIPTION:
An estimated total of 60 million people have been infected with HIV since the first cases were reported in the early 1980s. Although the HIV/AIDS pandemic is a global crisis, certain regions have been affected more than others. The Eastern European and Central Asian region, in particular, has one of the fastest growing rates of HIV infections in the world. Most new HIV infections in this region have been occurring among injection drug users, commercial sex workers, and men who have sex with men, but the virus continues to increasingly affect the general population, too. HIV prevention interventions that are able to be disseminated to a large population are necessary. The Popular Opinion Leader (POL) intervention is an HIV prevention program that recruits and trains opinion leaders in the community to promote safe sex behaviors through risk-reduction conversations with peers. Administering the POL intervention to nongovernmental organizations (NGOs) may be an effective means of assuring that the intervention is extended throughout the region. However, the best means of disseminating the POL program and assuring its full adoption by NGOs is unknown. This study will compare the effectiveness of face-to-face training versus Web-based training seminars in disseminating the POL intervention to NGOs in Eastern Europe and Central Asia.

Participation in this study will last 24 months. Potential NGOs will first undergo baseline assessments that will include an in-depth 90-minute phone interview with the NGO director and completion of attitude scales about the POL HIV intervention. NGOs will then be assigned randomly to one of three study groups:

* Participating NGOs in Group 1 will receive the POL intervention through face-to-face training. Staff will receive 2-day training on the POL intervention and individualized telephone follow-up consultations concerning POL implementation.
* Participating NGOs in Group 2 will receive the POL intervention through Web-based training. Staff will receive training delivered entirely by means of a Web-based, distance learning curriculum. Staff will also be offered individualized telephone follow-up consultations concerning POL implementation.
* Participating NGOs in Group 3 will receive no intervention.

All participating NGOs will undergo follow-up assessments 12 and 24 months after completing the intervention training. Assessments will include a 90-minute phone interview with the NGO director and a 10-minute phone interview with NGO staff members to assess attitudes concerning the intervention, their adoption of the core elements of the intervention model, and the extent of usage of training materials. A number of NGOs that report full adoption of the POL intervention will be selected randomly to undergo a 2-day validation site visit by an assessment team member. Site visits will be used to conduct interviews with NGO staff and the opinion leaders, validate reports of intervention adoption, observe POL sessions, and review materials used in training sessions.

ELIGIBILITY:
Inclusion Criteria for NGOs:

* Located in Eastern Europe or Central Asia
* Currently offers direct HIV prevention interventions targeting sexual risk in a community population
* Director willing to provide organizational consent
* Director and staff members willing to provide individual consent
* Director and staff members fluent in either English or Russian
* Has reliable Internet access

Exclusion Criteria for NGOs:

* Participated in prior Medical College of Wisconsin dissemination study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-11; Primary Completion 2013-02 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Adoption of the full Popular Opinion Leader intervention by a nongovernmental organization (NGO) | Measured at Months 12 and 24 after training

SECONDARY OUTCOMES:
Number of core elements of the Popular Opinion Leader intervention incorporated into NGO HIV prevention interventions | Measured at Months 12 and 24 after training
Cost effectiveness of training method | Measured at Month 24 after training

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin; Yuri A. Amirkhanian, PhD, Study Director — Medical College of Wisconsin; Timothy L. McAuliffe, PhD, Study Director — Medical College of Wisconsin; Laura R. Glasman, PhD, Study Director — Medical College of Wisconsin; Steven D. Pinkerton, PhD, Study Director — Medical College of Wisconsin
Locations (1):
- Center for AIDS Intervention Research, Medical College of Wisconsin, Milwaukee, Wisconsin, United States